CLINICAL TRIAL: NCT05328518
Title: Soft Tissue Tenderness and Fibromyalgia Among Schizophrenia Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Einat Mader, pricipal investigator, HaEmek Medical Center, Israel
Other Study IDs: 0052-20 EMC
Record Dates: First submitted 2022-03-14; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Fibromyalgia; Schizophrenia
MeSH Terms: conditions — Fibromyalgia; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Numerous studies reported on comorbidity of fibromyalgia and psychiatric disorders. Approximately 30% of patients with fibromyalgia have major depression at the time of diagnosis; the lifetime prevalence of depression is 74% and that of an anxiety disorder is 60%. In some fibromyalgia patients, mood and cognitive problems are much more prominent than tenderness. From the psychiatric point of view, 49% of PTSD patients and 5% of major depression patients fulfill criteria for diagnosing fibromyalgia.

The association between schizophrenia and fibromyalgia is still unknown.

Study hypothesis Schizophrenia patients, who have an aberrant sensation of pain, have lower prevalence of FM compared to the general population.

Primary objectives

1. Demonstrate that schizophrenia patients have lower prevalence of FM, compared to the general population.
2. To compare the self-reported extent and intensity of pain with selected tender points examination.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years of age.
* Patients must meet DSM-5 criteria for a diagnosis of schizophrenia.
* A stabled mental state.
* If hospitalized, patients are scheduled for discharge on the basis of clinical assessment of psychiatric symptoms.

Exclusion Criteria:

* Mental co-morbidity.
* Diagnosis of myofascial pain syndrome or chronic fatigue syndrome.
* Alcohol or drug use.
* Usage of any pain reliever medications during the week before recruitment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: schizophrenic womens
Sampling Method: Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
To compare the self-reported extent by questionnarie and intensity of pain with selected tender points examination. | 1 day
  To compare the self-reported extent and intensity of pain with selected tender points examination.
To compare between the degrees in pain recognition in schizophrenia patients who suffer from fibromyalgia to pain recognition in schizophrenia patients who do not suffer from fibromyalgia. | 1 day
  To compare between the degrees in pain recognition in schizophrenia patients who suffer from fibromyalgia to pain recognition in schizophrenia patients who do not suffer from fibromyalgia.

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel